CLINICAL TRIAL: NCT06505486
Title: Hepatic Arterial Infusion of GEMOX Plus Systemic Gemcitabine Chemotherapy Combined With Lenvatinib and PD-1 Inhibitor in Large Unresectable Intrahepatic Cholangiocarcinoma
Brief Title: GEMOX-HAIC Plus GEM-SYS in Combination With Lenvatinib and PD-1 Inhibitor for Large Unresectable ICC
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2024-539-01
Record Dates: First submitted 2024-07-11; First posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Intrahepatic Cholangiocarcinoma
Keywords: Intrahepatic Cholangiocarcinoma; Hepatic Arterial Infusion Chemotherapy; Immune Checkpoint Inhibitor; Tyrosine Kinase Inhibitor
MeSH Terms: conditions — Cholangiocarcinoma | interventions — gemcitabine-oxaliplatin regimen; lenvatinib; Immune Checkpoint Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HAIC+SYS+LEN+PD-1i
  Interventions: Drug: Gemcitabine-Oxaliplatin Regimen

INTERVENTIONS:
Drug: Gemcitabine-Oxaliplatin Regimen — Hepatic arterial infusion chemotherapy (HAIC) of gemcitabine and oxaliplatin (GEMOX) plus systemic gemcitabine chemotherapy (GEM-SYS) combined with lenvatinib and programmed cell death protein-1 (PD-1) inhibitor.
  Other Names: lenvatinib; PD-1 inhibitor

SUMMARY:
This study aimed to preliminarily evaluate the clinical efficacy and safety of hepatic arterial infusion chemotherapy (HAIC) of gemcitabine and oxaliplatin (GEMOX) plus systemic gemcitabine chemotherapy (GEM-SYS) combined with lenvatinib and programmed cell death protein-1 (PD-1) inhibitor in patients with large unresectable intrahepatic cholangiocarcinoma (uICC). Large uICC patients who underwent GEMOX-HAIC (Day 1) and GEM-SYS (Day 8) (3w/cycle) combined with lenvatinib and PD-1 inhibitor between November 2019 and December 2022 were enrolled. Clinical data were retrospectively collected to analyze local tumor response, progression-free survival (PFS), overall survival (OS), and adverse events (AEs). Tumor response was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. AEs were evaluated by the common terminology criteria for adverse events (CTCAE) version 5.0. In this study, OS was the primary endpoint, and progression-free survival (PFS) was the secondary endpoint.

ELIGIBILITY:
Inclusion Criteria:

(a) age of 18-70 years; (b) Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1; (c) diagnosis of ICC by histopathological examination of tissue biopsy specimens; (d) unresectable ICC confirmed by a multidisciplinary staff including at least one experienced liver surgeon; (e) tumor size larger than 5 cm in maximum diameter; (f) adequate liver function (total bilirubin < 3 times the upper limit of normal and aspartate/alanine transaminases < 5 times the upper limit of normal), adequate renal function (serum creatinine concentration of no more than 1.5 times the upper limit of the normal level), adequate bone marrow function (white blood cell count>3,000/mm3, hemoglobin>9.0g/dl and platelet count >100,000/mm3 ) and adequate coagulation function (prothrombin activity > 40% and international normalized ratio (INR) < 1.26); (g) patients received at least two cycles of GEMOX-HAIC + GEM-SYS combined with lenvatinib and PD-1 inhibitor; (h) patients with regular clinical data for evaluating the clinical efficacy and safety.

Exclusion Criteria:

(a) combined with other malignancies; (b) patients underwent any other chemotherapy regimens before, including gemcitabine and oxaliplatin; (c) patients received previous surgical resection or any other interventional procedures besides HAIC, such as transarterial chemoembolization (TACE), 125I seed implantation, radiofrequency ablation, microwave ablation, cryoablation, or percutaneous ethanol injection, etc.; (d) drug (chemotherapy drugs, lenvatinib, or PD-1 inhibitors) allergy; (e) patients with a history of autoimmune diseases; (f) patients with gastrointestinal bleeding of any grade within 4 weeks prior to the integrated treatment; (g) patients with uncontrolled comorbidities (e.g. general infection, serious dysfunction of heart or kidney, acute hepatitis or pneumonia, chronic obstructive pulmonary disease, or recent stroke).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 21 large uICC patients who underwent GEMOX-HAIC (Day 1) and GEM-SYS (Day 8) (3w/cycle) combined with lenvatinib and PD-1 inhibitor between November 2019 and December 2022 were enrolled.
Sampling Method: Probability Sample
Enrollment: 21 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2025-07-10 (Estimated); Study Completion 2025-07-10 (Estimated)

PRIMARY OUTCOMES:
Overall survival(OS) | 1-, 2-, and 3-year
  OS was calculated as the duration from the date of the first cycle of GEMOX-HAIC+GEM-SYS to the date of death or last date of follow-up.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 1-, 2-, and 3-year
  PFS was defined as the duration from the date of the first cycle of GEMOX-HAIC+GEM-SYS to tumor lesion progression, death, or last follow-up, whichever came first.

CONTACTS AND LOCATIONS:
Overall Officials: Jia-yan Ni, M.D., Principal Investigator — Sun Yat-sem Memorial Hospital, Sun Yat-sen University
Locations (1):
- Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University, Guangzhou, Guangzhou, China